CLINICAL TRIAL: NCT04128046
Title: The Effect of Platelet-rich Fibrin Matrix on Skin Rejuvenation: A Split Face Comparison
Brief Title: The Effect of Platelet-rich Fibrin Matrix on Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Manoj Abraham, Assistant Professor, New York Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12698
Record Dates: First submitted 2019-10-13; First posted 2019-10-16 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Skin Rejuvenation; Skin Quality; Wrinkle; Nasolabial Fold
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRFM (Experimental): Hemi-face injected with PRFM. PRFM was produced from 9 mL of blood (Healeon Medical, Inc).
  Interventions: Procedure: PRFM injection
- Saline (Placebo Comparator): Hemi-face injected with saline.
  Interventions: Procedure: Saline injection

INTERVENTIONS:
Procedure: PRFM injection — Using a 27-gauge microcannula, a total of 4 mL of PRFM was injected intradermally into the mid-cheek and NLF (2 mL for each site) on one side of the face.
  Arms: PRFM
Procedure: Saline injection — Using a 27-gauge microcannula, a total of 4 mL of saline was injected intradermally into the mid-cheek and NLF (2 mL for each site) on the contralateral side of the face.
  Arms: Saline

SUMMARY:
Platelet-rich fibrin matrix (PRFM) is made from platelets that are extracted from a patient's blood, and many plastic surgeons and dermatologists have used it to fill in wrinkles and lines on the face. Both patients and doctors have observed that it gives extra volume in these areas and improves overall appearance. However, there is no research that shows how PRFM affects skin quality, such as pores, spots, red areas, and texture. The aim of this study is to determine whether PRFM has a role in rejuvenating facial skin.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older who had a dermatological concern, specifically, conspicuous spots, pores, rhytids, uneven texture, or red or brown discoloration, and a VISIA complexion analysis score greater than 10
* Agreed to continue any contraceptive hormonal therapy for duration of the study
* Agreed to not initiate the use of hormonal therapy during the study
* Agreed to not undergo any facial procedures or treatments, including injections and fillers, lasers, peels, and topical therapies, during the duration of the study
* Agreed to adhere to a standardized skin care regimen throughout the duration of the study consisting of the use of a single cleanser and moisturizer twice a day
* Agreed to refrain from excessive sun exposure/tanning

Exclusion Criteria:

* History of skin/connective tissue disorders
* History of immunosuppressive therapy or radiotherapy
* Participation in facial procedures, such as injections, lasers, peels, and dermabrasion, in the last six months
* Use of topical/prescription acne medications in the last three months
* Current smokers or prior smokers who quit fewer than 10 years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in VISIA skin score | Skin analysis performed at initial visit, at 6 weeks, and at 12 weeks following initial treatment
  Difference between pre- and post-treatment VISIA analysis scores for skin parameters of spots, wrinkles, texture, and pores

SECONDARY OUTCOMES:
Change in Wrinkle Severity Rating Scale | Rating occurred at initial visit, at 6 weeks, and at 12 weeks following initial treatment
  Difference between pre- and post-treatment quantitative grading of nasolabial folds for each group. Graded from 1 through 5, with 5 representing the worst score
Skin Rejuvenation Outcomes Evaluation (SROE) | Evaluation distributed at initial visit, at 6 weeks, and at 12 weeks following treatment.
  Patient-reported outcome measure validated for skin resurfacing techniques. Each item is rated on a 0-4 scale. The final score is computed by dividing the total score for the instrument by 24 and multiplying by 100, giving a range of 0-100. The difference in the change in SROE score for each cohort was calculated.
VISIA Outcomes Questionnaire | Evaluation distributed at initial visit, at 6 weeks, and at 12 weeks following treatment.
  Evaluation targeted specifically at identifying changes in the skin parameters analyzed by VISIA. Each item is rated on a 0-4 scale. The final score is computed by dividing the total score for the instrument by 24 and multiplying by 100, giving a range of 0-100. The difference in the change in VISIA outcomes score for each cohort was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No